CLINICAL TRIAL: NCT01517763
Title: Comparison Study of the ICON™ Auto Series With and Without SensAwake™ and ThermoSmart™ and Conventional Continuous Positive Airway Pressure in Obstructive Sleep Apnea Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The site closed down, therefore the study has been terminated.
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: Sleep Health Centers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FPH-SA09-01
Record Dates: First submitted 2012-01-17; First posted 2012-01-25 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-05

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; Humidification; Continuous Positive Airway Pressure; ICON; ThermoSmart; SensAwake
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional CPAP (Placebo Comparator): Fisher & Paykel HC244™
  Interventions: Device: Conventional CPAP Therapy
- CPAP without Humidification (Active Comparator): Fixed pressure ICON™ without ThermoSmart™
  Interventions: Device: Fixed pressure ICON™ without ThermoSmart™
- APAP with all technologies (Experimental): Auto ICON™ with SensAwake™ and ThermoSmart™
  Interventions: Device: Auto ICON™ with SensAwake™ and ThermoSmart™

INTERVENTIONS:
Device: Conventional CPAP Therapy — HC244 devices without Thermosmart or SensAwake
  Arms: Conventional CPAP
Device: Fixed pressure ICON™ without ThermoSmart™ — Fixed pressure CPAP therapy using ICON™ without ThermoSmart™ or SensAwake™
  Arms: CPAP without Humidification
Device: Auto ICON™ with SensAwake™ and ThermoSmart™ — APAP therapy using Auto ICON™ with SensAwake™ and ThermoSmart™
  Arms: APAP with all technologies

SUMMARY:
A total of 216 patients will be randomized into a partially single blind, randomized, parallel-arm trial to determine whether the ICON™ AT with SensAwake™ and ThermoSmart™ can improve therapy adherence when compared to standard care with a fixed pressure Continuous Positive Airway Pressure (CPAP) device and compared to a less aesthetically pleasing CPAP device without technologies (AutoCPAP, SensAwake™, ThermoSmart™) in patients previously diagnosed with moderate-severe obstructive sleep apnea (OSA).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years with moderate-to-severe OSA (Apnea Hypopnea Index equal to or greater than 10 per hour).
* Successful titration Polysomnography (PSG).
* Fluency in both written and spoken English.

Exclusion Criteria:

* Participants prescribed and fitted with any PAP device in the past 2 years.
* Contraindicated for CPAP or AutoCPAP therapy.
* Any known factor or disease that might interfere with treatment adherence, study conduct or interpretation of the results such as severe psychiatric disease, history of non adherence to medical regimens, or unwillingness to comply with study requirements as determined by the principal investigator.
* Other significant sleep disorder(s) that would interfere with their ability to wear CPAP as determined by the principal investigator.
* Previous surgery for OSA or snoring or any surgery of the mouth, nose, sinuses or airways.
* If SensAwake™ or ThermoSmart™ was disabled on the treatment arm (or conversely) during the study protocol.
* If participants are required, by the nature of their employment, to comply with therapy. For example truck drivers or airline pilots.
* If the physician objects to their patient taking part in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep HealthCenters, Brighton, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This trial was terminated due to abrupt and unexpected closure of all study sites. All case report forms and consent forms were lost as a result and therefore, there are no results to report as no data exists.
Period: Overall Study
Arm/Group | Conventional CPAP | CPAP Without Humidification | APAP With All Technologies
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This trial was terminated due to abrupt and unexpected closure of all study sites. All case report forms and consent forms were lost as a result and therefore, there are no results to report as no data exists.
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional CPAP | CPAP Without Humidification | APAP With All Technologies | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Adherence With Treatment Per Night Averaged Over Total Time Period Measured Via Internal Software on the Device and Reported on Using InfoSmart™ Software.
Time Frame: On day 90 after randomization
Population: as for baseline characteristics
Arm/Group | Conventional CPAP | CPAP Without Humidification | APAP With All Technologies
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Adherence (Hours of Usage Per Night) and Acceptance (Number of Drop-outs). Complaints During Follow up Calls and Visit.
Time Frame: On day 90 after randomization
Population: as for baseline characteristics
Arm/Group | Conventional CPAP | CPAP Without Humidification | APAP With All Technologies
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: This trial was terminated due to abrupt and unexpected closure of all study sites. All case report forms and consent forms were lost as a result and therefore, there are no results to report as no data exists.
Arm/Group | Conventional CPAP | CPAP Without Humidification | APAP With All Technologies
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This trial was terminated due to abrupt and unexpected closure of all study sites. All case report forms and consent forms were lost as a result and therefore, there are no results to report as no data exists.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No